CLINICAL TRIAL: NCT06392802
Title: Effectiveness of a Rehabilitation Exercise Plan at Home to Treat Post-stroke Patients in the Chronic Phase
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Politècnica de Catalunya (Other)
Collaborators: Consorci Hospitalari de Vic (Other); Institut Català de la Salut (Other); EAP Vic (CAP Remei) (Unknown); Associació Disminuïts Físics d'Osona (Unknown)
Responsible Party: Principal Investigator, Gil Serrancolí, Principal Investigator, Universitat Politècnica de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RehabAtHome_Osona
Record Dates: First submitted 2024-01-17; First posted 2024-04-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Motor Disorders; Physical Disability
Keywords: post-stroke; telerehabilitation; non-immersive virtual reality
MeSH Terms: conditions — Stroke; Motor Disorders

STUDY DESIGN:
Intervention Model Description: Two groups of 25 subjects follow a motor rehabilitation treatment during 12 weeks. One group (Control group) uses the typical rehabilitation process (just doing exercises at home, written on a sheet of paper). The intervention group uses the telerehabilitation system Muvity during 12 weeks at home to perform motor exercises and play exergames.
Who Masked: Care Provider, Investigator
Masking Description: Both groups are assessed by a blinded physiotherapist, before and after the treatments. This does not know in which group the participant is involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group follows a treatment similar to the one that a public hospital recommends. They receive a sheet of paper with the description of some exercises to do at home. These should be done in three 30-min-sessions per week, during 12 weeks.
- Muvity - Intervention (Experimental): This group follows a treatment prescribed by a therapist using Muvity, a telerehabilitation system using a depth camera. The treatment consists of some exercises guided by a virtual avatar, and some exergames to play. The computer application monitors the ranges of motion of joint angles as well as time played and deviations from theoretical trajectories. These sessions are programmed to be done in three 30-min-sessions per week, during 12 weeks (same amount as the Control group).
  Interventions: Device: Rehabilitation treatment using Muvity

INTERVENTIONS:
Device: Rehabilitation treatment using Muvity — The users have the support of the telerehabilitation system Muvity
  Arms: Muvity - Intervention

SUMMARY:
Background: Stroke is the second leading cause of death worldwide and the primary medical cause of disability. It is estimated that 45% of affected individuals will continue to have moderate or severe functional disabilities throughout their lives. According to the American Stroke Association, telerehabilitation has the potential to provide timely and efficient care to stroke survivors, improving patients' functional outcomes while reducing long-term disability and associated costs.

Hypothesis: Through the developed application (Muvity), the study aims to contribute to the validity of telerehabilitation and virtual reality as beneficial tools for rehabilitation, specifically for individuals in the post-stroke sequelae phase.

Objectives: To evaluate the effectiveness of a non-immersive virtual reality program in telerehabilitation for patients who have experienced a stroke more than 6 months ago.

Methodology: Prospective longitudinal study with single blinding. The control group undergoes a conventional intervention, while the experimental group undergoes an innovative intervention (n=25).

Variables: The collected variables and measurement tools include upper extremity functionality (Fugl-Meyer scale), balance (Berg), functional independence (Barthel), pain (Brief Pain Inventory), post-stroke quality of life (ECVI-38), emotional health (UCLA Self-Rating Depression Scale), treatment expectations (Expectation for Treatment Scale), treatment adherence (through an APP), and satisfaction (Telehealth Usability Questionnaire).

Statistical Analysis: Data will be analyzed per protocol (PP); the normality distribution of the data will be assessed, and results will be analyzed using parametric or non-parametric techniques depending on normality. A bivariate analysis will compare results between the control and intervention groups, considering a statistically significant result when p < 0.05.

Expected Results: Similar results are expected between groups or slightly favorable outcomes in the experimental group for the different variables.

Applicability and Relevance: The application would facilitate access to motor rehabilitation treatments in an enjoyable and engaging manner, promoting physical activity and contributing to a healthy lifestyle. Upon obtaining the results of this study, a trial implementation of the application in five socio-sanitary or associative centers is planned to verify its final applicability.

DETAILED DESCRIPTION:
As described in the "Catalan Consensus on Evaluation and Treatment of Post-Stroke Patients," in the chronic phase when the effects of stroke have stabilized, patients should continue to have access to rehabilitation services to address their long-term needs. However, the decision to refer patients to rehabilitation services often relies heavily on patient and family demand, lacking clear criteria to ensure coordination between Primary Care services and specialized ones. Considering this gap in action, along with the estimated high costs associated with caring for stroke survivors, non-immersive virtual reality telerehabilitation is proposed as a beneficial tool for both patients and healthcare professionals and managers.

The study aims to contribute to the validity of telerehabilitation and virtual reality as beneficial tools for rehabilitation, specifically for individuals experiencing post-stroke sequelae.

Objectives (General and Specific)

The general objective of this study is to evaluate the effectiveness of a non-immersive virtual reality program in telerehabilitation targeting subjects who have suffered a stroke for more than six months, comparing the effectiveness of conventional therapy with gamified therapy (using the developed computational application).

The specific objectives of the study are as follows:

* Observe changes in joint range of motion (flexion, abduction, horizontal abduction of the shoulder, and elbow flexion) before and after the intervention.
* Assess if game performance (scores, time, etc.) changes between week 2 and week 12.
* Analyze the effects of the computational application on users' balance. Compare balance results between both groups.
* Measure the evolution of the pain variable before and after the intervention and compare it between the two groups.
* Explore potential changes in users' emotional health throughout the intervention.
* Determine the impact of the application on the user's quality of life (QoL).
* Verify if subjects' expectations are met through the application's use.
* Compare treatment adherence using the application versus conventional methodology.
* Determine if using the application leads to greater satisfaction in offering home rehabilitation guidance.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 85 years old.
* Stroke duration of more than six months + Discharge from post-stroke rehabilitation.
* Moderate physical disability: scoring between 1-3 on the Modified Rankin Scale.
* Standing: able to stand safely for 2 minutes without support (maximum score -4- on item 2 of the Berg Scale).
* Vision: capable of correctly visualizing a screen at a distance of 2 meters.
* Cognitive status: No cognitive impairment or mild cognitive impairment (Mini-Mental State Examination score ≥ 24). Ability to understand and follow verbal instructions in Catalan or Spanish.
* Technological skills: capable of basic use of a mobile phone and computer (keyboard, mouse, screen).
* Glenohumeral joint mobility: minimum of 30º flexion, abduction, horizontal abduction; and 15º internal and external rotation.
* Elbow joint mobility: minimum of 45º flexion.

Exclusion Criteria:

* Engaging in intense physical therapies.
* Severe aphasia: inability or difficulty communicating through speech.
* Cognitive impairments affecting short and mid-term memory.
* Vision: having visual deficits in either eye that may impair screen visualization.
* Vision: experiencing hemispatial neglect, meaning difficulty processing stimuli on the side opposite to the injury.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, female, non-binary
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer | Within one week before and within one week after the treatments for both groups.
  Standard Fugl-Meyer score to assess motor functionality. Sections A (upper limbs, up to 36 points), D (coordination, up to 6 points), H (sensation, up to 6 points), I (joint movement (up to 16 points), and J (joint pain, up to 16 points). The total score could be up to 80 points (the higher score, the higher functionality).
Berg score | Within one week before and within one week after the treatments for both groups.
  The Standard Berg Balance Scale is used to assess balance control. Scores range from 0 (equilibrium heavily affected) to 56 (excellent equilibrium capacity).
Brief Pain Inventory | Within one week before and within one week after the treatments for both groups.
  Standard score to assess joint pain. It consists of 11 questions related to pain intensity. A score of 0 indicates pain absence, and 10 high pain intensity.
Ranges of motion | Within one week before and within one week after the treatment for both groups and during the 12-week treatment for the intervention group.
  The ranges of motion of upper and lower limb joint angles are computed before and after the treatments for both control and intervention groups during the assessment face-to-face sessions. This information is also gathered for the intervention group during the 12-week treatment.

SECONDARY OUTCOMES:
Ranges of motion | During the 12-week treatment for the intervention group.
  The ranges of motion of upper and lower limb joint angles are computed before and after the treatments for both control and intervention groups during the assessment face-to-face sessions. This information is also gathered for the intervention group during the 12-week treatment
Time spent for the rehabilitation sessions | During the 12-week treatment for the intervention group.
  The time spent for the rehabilitation sessions is monitored for both groups (by a simple mobile app for the Control group and by Muvity for the intervention group)
ECVI-38 | Within one week before and within one week after the 12-week treatment
  Quality of life is monitored by the standard test ECVI-38. This stands for "Escala de calidad de vida para el ictus" (ECVI) in Spanish (Quality of Life Scale for Stroke), It ranges between 0 (no impairment) to 100 (maximum impairment).
UCLA Self-Rating Depression Scale | Within one week before and within one week after the 12-week treatment
  Self-rating depression score. It ranges between 3 (low perception of loneliness) to 9 (high perception of loneliness).

CONTACTS AND LOCATIONS:
Overall Officials: Gil Serrancolí, PhD, Principal Investigator — Universitat Politècnica de Catalunya; Cris Molas, Msc, Principal Investigator — Associació Disminuïts Físics d'Osona
Locations (2):
- Spain (2):
  - Associació Disminuïts Físics d'Osona, Vic, Barcelona
  - Universitat Politècnica de Catalunya, Barcelona

IPD SHARING:
Plan to Share IPD: No
We aim to disseminate the aggregated results. The identification of each participant will not be possible for the researchers who will use these data.